CLINICAL TRIAL: NCT00776256
Title: The Effect of Meal Replacement Bars Containing Different Types of Fibres (Oligofructose and/or Barley) on Satiety and Energy Intake
Brief Title: Effects of Oligofructose and Barley on Satiety and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Harry Peters, Unilever R&D
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 07002V
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Appetite Regulation
Keywords: satiety; food intake
MeSH Terms: interventions — beta-Glucans; fructooligosaccharide; oligofructose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): effect of beta-glucan
  Interventions: Dietary Supplement: beta-glucan and fructooligosaccharide
- 2 (Active Comparator): effect of fructo-oligosaccharide
  Interventions: Dietary Supplement: beta-glucan and fructooligosaccharide
- 3 (Active Comparator): effect of beta-glucan and fructooligosaccharide
  Interventions: Dietary Supplement: beta-glucan and fructooligosaccharide
- 4 (Placebo Comparator): no beta-glucan nor fructooligosaccharide
  Interventions: Dietary Supplement: beta-glucan and fructooligosaccharide

INTERVENTIONS:
Dietary Supplement: beta-glucan and fructooligosaccharide — 1g beta-glucan or 8 g fructooligosaccharide or combination per meal replacement bar given twice on day 1 and once on day 2
  Other Names: oats; barley; oligofructose

SUMMARY:
The effect of beta-glucan or fructo-oligosaccharide or their combination in bars on satiety and food intake was tested by supplying these bars on two consecutive days.

DETAILED DESCRIPTION:
Background: Increasing gastro-intestinal viscosity or colonic fermentation is suggested to help improve appetite control and reduce food intake. Beta-glucan (BG) and fructo-oligosaccharide (FOS) are food ingredients proposed to act this way, but results so far remain inconclusive.

Objective: To test the effect of FOS, BG, or their combination in bars on appetite ratings and food intake during 2 consecutive days.

Design: In a 4-way balanced order cross-over double-blind design, 21 healthy volunteers (mean BMI 25.9 kg/m2) received a meal replacement bar at 09.00h and an ad libitum lunch at 13.00h on 2 consecutive days. On day 1 only, subjects consumed a second (identical) bar at 17.00h and a fixed snack at 19.00h. The control bar contained 0.3g BG (control, from 6.8 g oats), vs equi-caloric bar formulations containing an additional: 1) 0.9 g BG (from 8.0g barley), 2) 8g FOS, or 3) 0.9 g BG + 8g FOS. Appetite scores and subsequent ad libitum test meal intakes were measured. Bar viscosities were determined under simulated gastric conditions. Results were analyzed using ANCOVA.

Results: Addition of BG, FOS or their combination did not affect appetite ratings or food intake, although addition of BG to the bar doubled apparent gastric viscosity (841 vs 351 mPa.s).

Conclusions: BG, FOS or their combination in bars at these levels do not improve appetite control when consumed on 2 consecutive days. Efficacy might be increased by a longer exposure period, increasing the BG content, or a form of BG that generates even higher gastric viscosity.

ELIGIBILITY:
Inclusion Criteria:

* Age at start of the study 18 till 60 years
* Quetelet-Index (BMI) from 21 till 32 kg/m2 inclusive
* Apparently healthy: measured by questionnaire: no reported current or previous metabolic diseases or chronic gastrointestinal disorders
* Reported dietary habits: no medically prescribed diet, no slimming diet, used to eat 3 meals a day, no vegetarian, macro-biotic or biologic dynamic food habits
* No Fibre supplements (only once a day)
* No blood donations during the study.
* Reported intense sporting activities less than 10h/w
* Reported alcohol consumption less than 21 units/w (female volunteers) or less than 28 units/w (male volunteers)
* Having a General Practitioner
* Informed consent signed
* Recruitment form filled out

Exclusion Criteria:

* Smoking
* Dislike, allergy/intolerance or not known with the foods of the ad libitum meal
* Possible eating disorder (measured by SCOFF questionnaire)
* High or very high restrained eaters (measured by questionnaire) (men with BMI < 27: restraint score > 2.37, men with BMI less than 27: restraint score > 3.04, women with BMI < 26: restraint score > 3.24, women with BMI less than 26: restraint score > 3.41)
* Reported medical treatment that may affect eating habits/satiety
* Reported intolerance or allergy to test products
* Women reported lactating (or lactating < 6 weeks ago), pregnant (or pregnant < 3 months ago) or wish to become pregnant during the study
* Reported weight loss/gain (10%) in the last six month before the trial
* Reported participation in another biomedical trial 1 month before the start of the study
* Reported working on late turns -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Satiety and food intake | 2 days each week for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward Haddeman, Study Director — Unilever R&D
Locations (1):
- Unilever R&D Vlaardingen, Vlaardingen, Netherlands

REFERENCES:
- [Derived] Peters HP, Boers HM, Haddeman E, Melnikov SM, Qvyjt F. No effect of added beta-glucan or of fructooligosaccharide on appetite or energy intake. Am J Clin Nutr. 2009 Jan;89(1):58-63. doi: 10.3945/ajcn.2008.26701. Epub 2008 Dec 3. PMID 19056555